CLINICAL TRIAL: NCT01668095
Title: Developmental Pathway Drug-Targets in Advanced Rhabdomyosarcomas
Brief Title: Biomarkers in Patients With Advanced Rhabdomyosarcoma
Status: Completed | Type: Observational
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: ARST12B8; NCI-2012-01997 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); COG-ARST12B8 (Other: Children's Oncology Group); CDR0000738499 (Other: Clinical Trials.gov); ARST12B8 (Other: Children's Oncology Group); ARST12B8 (Other: CTEP)
Record Dates: First submitted 2012-08-15; First posted 2012-08-17 (Estimated); Last update posted 2016-05-18 (Estimated); Status verified 2016-05

CONDITIONS: Adult Rhabdomyosarcoma; Childhood Alveolar Rhabdomyosarcoma; Childhood Embryonal Rhabdomyosarcoma; Previously Treated Childhood Rhabdomyosarcoma; Recurrent Adult Soft Tissue Sarcoma; Recurrent Childhood Rhabdomyosarcoma; Stage III Adult Soft Tissue Sarcoma; Stage IV Adult Soft Tissue Sarcoma
MeSH Terms: conditions — Rhabdomyosarcoma; Sarcoma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — tumor tissue
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Ancillary-Correlative (biomarker analysis): Immunohistochemistry is performed for each candidate target (Pax3, Pax7, and Patched-1) in each disease (alveolar, embryonal, and anaplastic rhabdomyosarcoma) for tissue microarray analysis.
  Interventions: Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Other: Laboratory Biomarker Analysis — Correlative studies

SUMMARY:
This research trial studies tumor tissue to identify important proteins and biomarkers from patients with rhabdomyosarcoma that has spread to other places in the body and usually cannot be cured or controlled with treatment. Studying samples of tumor tissue from patients with cancer in the laboratory may help doctors identify biomarkers related to cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To investigate whether the expression of a subset of proteins (by immunohistochemistry), known to be Involved in the paired box (Pax)3, Pax7, and Patched-1 neuromuscular development pathways, are dysregulated in advanced and relapsed alveolar and embryonal rhabdomyosarcomas.

OUTLINE:

Immunohistochemistry is performed for each candidate target (Pax3, Pax7, and Patched-1) in each disease (alveolar, embryonal, and anaplastic rhabdomyosarcoma) for tissue microarray analysis.

ELIGIBILITY:
Inclusion Criteria:

* 8 tissue microarrays (TMA) slides of the following diseases available:

  * Alveolar rhabdomyosarcoma
  * Embryonal rhabdomyosarcoma
  * Anaplastic rhabdomyosarcoma

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with rhabdomyosarcoma that has spread to other places in the body and usually cannot be cured or controlled with treatment.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2012-08; Primary Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Prevalence of the candidate target (Pax3, Pax7, or Patched-1), and whether the candidate target is expressed in the tumor vs stroma | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Charles Keller, MD, Principal Investigator — Children's Oncology Group
Locations (1):
- Children's Oncology Group, Philadelphia, Pennsylvania, United States